CLINICAL TRIAL: NCT01570777
Title: Renal Denervation in Patients With Resistant Hypertension
Brief Title: Renal Denervation in Hypertension
Acronym: DENER-HTN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110127
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Hypertension, Resistant to Conventional Therapy; Renal Denervation
Keywords: Resistant hypertension; Renal denervation; Standardized medication regimen; Endovascular; Primary hypertension; Cardiovascular diseases; Vascular diseases
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Essential Hypertension; Cardiovascular Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal denervation (Experimental)
  Interventions: Procedure: renal denervation and optimized medication regimen
- optimized medication regimen (Other): optimized medication regimen
  Interventions: Procedure: optimized medication regimen

INTERVENTIONS:
Procedure: renal denervation and optimized medication regimen — Patients are treated with the renal denervation plus a standardized optimal antihypertensive treatment which is adapted every month starting two month after randomization on the basis of home BP monitoring results at follow-up visits.
  Other Names: TMAOS + DR
  Arms: Renal denervation
Procedure: optimized medication regimen — Patients are treated with a standardized optimal antihypertensive treatment which is adapted every month starting two month after randomization on the basis of home BP monitoring results at follow-up visits.
  Other Names: TMAOS
  Arms: optimized medication regimen

SUMMARY:
The DENER-HTN study is a, multicenter, prospective, open, randomized, controlled study of the effectiveness and costs of renal denervation in addition to standardized medical treatment compared to medical treatment alone in subjects with resistant hypertension. Bilateral renal denervation will be performed using the Symplicity Catheter - a percutaneous system that delivers radiofrequency (RF) energy through the luminal surface of the renal artery.

DETAILED DESCRIPTION:
The DENER-HTN study is a, multicenter, prospective, open, randomized, controlled study of the efficacy and cost-effectiveness of renal denervation plus standardized optimal antihypertensive treatment compared to standardized optimal antihypertensive treatment alone in patients with proven resistant hypertension. Patients with essential resistant hypertension will first enter a 4-week run-in period during which they will receive a standardized triple combination therapy (diuretic+ ACE inhibitor+ CCB at maximal dose). After 4 weeks of standardized triple therapy patients will be randomized to renal denervation + optimal antihypertensive treatment compared to standardized optimal antihypertensive treatment if daytime ambulatory BP remains ≥ 135 and/or 85 mmHg. Bilateral renal denervation will be performed using the Symplicity Catheter (Medtronic ®) - a percutaneous system that delivers radiofrequency (RF) energy through the luminal surface of the renal artery. Study amendment: Extended follow-up of 48 months for all randomized patients.

ELIGIBILITY:
Inclusion Criteria:

* Individual is more than 18 and less than 75 years old at time of randomization
* Essential hypertension diagnosed during a complete work-up within the past 2 years
* Office blood pressure ≥140 and/or 90 mmHg despite a stable medication regimen including full tolerated doses of 3 or more anti-hypertensive medications of different classes, including a diuretic
* 2 functional kidneys sizing ≥ 90 mm; eGFR ≥ 40 mL/min/1.73m² (MDRD formula)
* Suitable renal anatomy compatible with the endovascular denervation procedure
* Signed Informed consent
* Confirmed resistant hypertension defined by diurnal ambulatory blood pressure measurement ≥ 135 and/or 85 mmHg after 4 week standardized triple antihypertensive treatment

Exclusion Criteria:

* Patients with an estimated glomerular filtration rate (eGFR) of less than 40 mL/min/1.73 m2
* Patients with secondary hypertension
* Kaliemia ≥ 6mmol/L
* Patient with single functioning kidney
* Patient with contrast media allergy
* Patient with any implantable device incompatible with radiofrequency energy delivery
* Patient with contra-indication to the anti-hypertensive standardized medication regimen
* Patient with transient or fixed cerebral ischemia within 3 months before inclusion
* Patient with myocardial infarction, unstable angina pectoris, coronary bypass or percutaneous angioplasty within 3 months before inclusion
* Patient with type 1 diabetes mellitus
* Patient with malignancy within the 5 past years
* Patient with atrial fibrillation and/or a brachial circumference of ≥ 42cm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Mean diurnal systolic blood pressure assessed by ABPM | Baseline to 6 months
Cost-effectiveness evaluation | 1 year

SECONDARY OUTCOMES:
Antihypertensive medication score | baseline to 15 months
Adverse events of renal denervation | baseline to 48 months
Detailed analysis of blood pressure | baseline to 15 months
Change in average 24-hour and nighttime Systolic Blood Pressure by ambulatory blood pressure monitoring | baseline to 15 months
Change in average 24-hour, daytime and nighttime diastolic Blood Pressure, pulse pressure and heart rate by ambulatory blood pressure monitoring | baseline to 15 months
Change in Systolic/diastolic Blood Pressure by home blood pressure monitoring | baseline to 15 months
Change in office Systolic/diastolic Blood Pressure | baseline to 15 months
Adherence to antihypertensive Medication | baseline to 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc SAPOVAL, PD, PhD, Principal Investigator — departement of interventional radiology
Locations (1):
- CIC Hopital europeen george pompidou, Paris, France

REFERENCES:
- [Derived] Hamdidouche I, Gosse P, Cremer A, Lorthioir A, Delsart P, Courand PY, Denolle T, Halimi JM, Girerd X, Ormezzano O, Rossignol P, Pereira H, Azizi M; DENERHTN Investigators. Clinic Versus Ambulatory Blood Pressure in Resistant Hypertension: Impact of Antihypertensive Medication Nonadherence: A Post Hoc Analysis the DENERHTN Study. Hypertension. 2019 Nov;74(5):1096-1103. doi: 10.1161/HYPERTENSIONAHA.119.13520. Epub 2019 Sep 23. PMID 31995406
- [Derived] Courand PY, Pereira H, Del Giudice C, Gosse P, Monge M, Bobrie G, Delsart P, Mounier-Vehier C, Lantelme P, Denolle T, Dourmap C, Halimi JM, Girerd X, Rossignol P, Zannad F, Ormezzano O, Vaisse B, Herpin D, Ribstein J, Bouhanick B, Mourad JJ, Ferrari E, Chatellier G, Sapoval M, Azarine A, Azizi M; DENERHTN Investigators. Abdominal Aortic Calcifications Influences the Systemic and Renal Hemodynamic Response to Renal Denervation in the DENERHTN (Renal Denervation for Hypertension) Trial. J Am Heart Assoc. 2017 Oct 10;6(10):e007062. doi: 10.1161/JAHA.117.007062. PMID 29018027
- [Derived] Gosse P, Cremer A, Pereira H, Bobrie G, Chatellier G, Chamontin B, Courand PY, Delsart P, Denolle T, Dourmap C, Ferrari E, Girerd X, Michel Halimi J, Herpin D, Lantelme P, Monge M, Mounier-Vehier C, Mourad JJ, Ormezzano O, Ribstein J, Rossignol P, Sapoval M, Vaisse B, Zannad F, Azizi M. Twenty-Four-Hour Blood Pressure Monitoring to Predict and Assess Impact of Renal Denervation: The DENERHTN Study (Renal Denervation for Hypertension). Hypertension. 2017 Mar;69(3):494-500. doi: 10.1161/HYPERTENSIONAHA.116.08448. Epub 2017 Jan 23. PMID 28115517
- [Derived] Azizi M, Pereira H, Hamdidouche I, Gosse P, Monge M, Bobrie G, Delsart P, Mounier-Vehier C, Courand PY, Lantelme P, Denolle T, Dourmap-Collas C, Girerd X, Michel Halimi J, Zannad F, Ormezzano O, Vaisse B, Herpin D, Ribstein J, Chamontin B, Mourad JJ, Ferrari E, Plouin PF, Jullien V, Sapoval M, Chatellier G; DENERHTN Investigators. Adherence to Antihypertensive Treatment and the Blood Pressure-Lowering Effects of Renal Denervation in the Renal Denervation for Hypertension (DENERHTN) Trial. Circulation. 2016 Sep 20;134(12):847-57. doi: 10.1161/CIRCULATIONAHA.116.022922. Epub 2016 Aug 30. PMID 27576780
- [Derived] Azizi M, Sapoval M, Gosse P, Monge M, Bobrie G, Delsart P, Midulla M, Mounier-Vehier C, Courand PY, Lantelme P, Denolle T, Dourmap-Collas C, Trillaud H, Pereira H, Plouin PF, Chatellier G; Renal Denervation for Hypertension (DENERHTN) investigators. Optimum and stepped care standardised antihypertensive treatment with or without renal denervation for resistant hypertension (DENERHTN): a multicentre, open-label, randomised controlled trial. Lancet. 2015 May 16;385(9981):1957-65. doi: 10.1016/S0140-6736(14)61942-5. Epub 2015 Jan 26. PMID 25631070
- [Derived] Persu A, Sapoval M, Azizi M, Monge M, Danse E, Hammer F, Renkin J. Renal artery stenosis following renal denervation: a matter of concern. J Hypertens. 2014 Oct;32(10):2101-5. doi: 10.1097/HJH.0000000000000323. No abstract available. PMID 25186534